CLINICAL TRIAL: NCT02066311
Title: Nelfinavir in Systemic Lupus Erythematosus: A Pilot Phase IIa Clinical Trial
Brief Title: Nelfinavir in Systemic Lupus Erythematosus
Acronym: NISLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stage 1 terminated 6/1/18 prior to completion of Stage 1 due to low enrollment and efficacy
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Meggan Mackay, Associate Investigator, MD, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NISLE
Record Dates: First submitted 2014-02-12; First posted 2014-02-19 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nelfinavir (Experimental): Nelfinavir tablets will be taken by oral administration, 750mg (three 250 mg tablets) three times a day
  Interventions: Drug: Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir
  Other Names: Viracept

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune disease in which the body's immune system attacks different parts of the body. SLE is characterized by inflammation that leads to tissue damage in different organ systems. Any organ system may be involved, including the skin, the joints, the kidneys, the nervous system, the heart, the lungs, and the blood. The exact cause of SLE is not known. Patients with SLE often have elevated levels of anti-double stranded DNA antibodies. These levels are often associated with disease flares and disease severity. These antibodies can bind to tissue leading to organ damage. Preventing these antibodies from binding to their targets may help decrease disease activity.

Protease inhibitors are medications that have been approved by the Food and Drug Administration (FDA) for use in the treatment of HIV (human immunodeficiency virus). Nelfinavir (also called viracept) is one of these protease inhibitors. Separate from their anti-viral effects, protease inhibitors have been found to decrease inflammation. These medications have been shown to interfere with binding of anti-double stranded DNA antibodies to their targets and may decrease inflammation in SLE. This research study tests whether the protease inhibitor, nelfinavir, will decrease anti-double stranded DNA antibody binding and decrease disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is capable of providing written informed consent
2. Subject is ≥ 18 years old and ≤ 65 years old
3. Meets at least 4 of 11 modified American College of Rheumatology (ACR) (1997) Revised Criteria for the Classification of Systemic Lupus Erythematosus
4. Has mild to moderate disease activity defined as

   * A minimum SLEDAI score of 2 excluding points for serology (anti-dsDNA antibody and complement)
   * No active renal or nervous system disease
   * No BILAG A in any organ system
   * No expectation by the investigator that corticosteroids will need to be added or doses increased during the 8 week treatment period for any reason
   * No expectation by the investigator that immunosuppressive medication will need to be added or doses increased during the 8 week treatment period
5. Has elevated titers of anti-ds DNA antibody at the time of screening (defined as the titer that meets criteria for "high" in the Core Laboratory at the North Shore/LIJ Health Systems; unequivocal high titer as opposed to borderline, indeterminate or intermediate).
6. Has elevated titers of cross-reactive anti-DNA/DWEYS antibodies at the time of screening (the assays for anti-DNA/DWEYS antibodies will be performed in Dr. B. Diamond's laboratory; study sites will be notified of results within 3 days of receipt of the samples).
7. If on glucocorticoids, the dose must be ≤10 mg daily and stable for the 4 weeks prior to screening and baseline
8. If on immunosuppressive or immunomodulatory medication such as azathioprine, methotrexate, leflunomide, mycophenolate, or hydroxychloroquine, the dose must have been stable for the 3 months prior to screening, and expected to remain stable over the course of the study.
9. Males and females with potential for reproduction must agree to practice effective birth control measures (2 approved methods of contraception). Nelfinavir can decrease serum levels of oral contraceptives; the slightly increased risk of pregnancy due to an interaction between oral contraception and nelfinavir will be discussed when appropriate and the requirement for a second approved method of contraception will be addressed.

Exclusion Criteria:

1. Current or prior treatment with rituximab, belimumab or anti-CD22 monoclonal antibody in the 12 months prior to this study or any other biologic agent for 90 days prior to this study
2. Treatment with cyclophosphamide within the 6 months prior to screening
3. Increase in glucocorticoid dose within 4 weeks of screening or addition of a DMARD in the three months prior to study
4. A history of drug or alcohol abuse within the 6 months prior to screening
5. Elevated LFT's:

   * ALT or AST ≥ 2 x upper limit of normal at screening
   * serum unconjugated bilirubin > 3mg/dL at screening
6. Dialysis or serum creatinine >1.5mg/dL
7. Hypercholesterolemia: total cholesterol >230 mg/dL or LDL >150 mg/dl or hypertriglyceridemia (triglyceride >200mg/dL) at screening
8. Laboratory/clinical evidence of: pancreatitis: amylase/lipase >3x upper limit of normal at screening
9. Known current/active infections including HIV, Hepatitis B, Hepatitis C
10. History of cancer, excluding skin cancers (squamous cell or basal cell that have been treated)
11. Known active tuberculosis or untreated tuberculosis
12. Hemoglobin < 8 g/dL
13. Expectation by the investigator to increase corticosteroid or immunosuppressive, or immunomodulatory medication dose at screening, baseline, or over the course of the study
14. Pregnancy or lactation
15. Consumption of > 2 cups of grapefruit juice per day
16. Treatment with medications metabolized using the cytochrome P3A4 pathway, such as cyclosporine, tacrolimus, gemfibrozil, niacin, itraconazole, ketoconazole, erythromycin, azithromycin, clarithromycin, bosentan, nefazodone, tricyclic antidepressants
17. Any condition that, in the opinion of the Investigator, would jeopardize the subject's safety following exposure to the study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meggan Mackay, MD, Principal Investigator — Northwell Health
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - New York University School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Bronx Lebanon Hospital, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Study With the Simon Two-Stage Trial Design: All subjects will be dosed with nelfinavir 750 mg orally three times daily. This dose may be decreased to 750 mg twice daily if not tolerated. For both stages of the trial the dosing period is 8 weeks followed by a 4 week observation period.
  A maximum of 13 subjects will be enrolled in Stage 1. From the 13 subjects enrolled in Stage 1; if 3 or fewer subjects achieve a Response (a ≥35% reduction in serum anti-dsDNA antibody titer), the trial will be terminated. If 4 or more subjects achieve a Response, the study will be expanded to enroll an additional maximum of 30 patients in Stage 2.
Period: Overall Study
Arm/Group | Open-label Study With the Simon Two-Stage Trial Design
Started | 15
Completed | 10 (Stage 1 terminated 6/1/18 prior to completion of Stage 1 due to low enrollment and efficacy.)
Not Completed | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Study With the Simon Two-Stage Trial Design
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 15
Serum anti-dsDNA antibody titer [Mean (Standard Deviation); unit: IU/mL] | 313.8 (299.7)

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of Anti-dsDNA Binding
Description: Change in serum anti-dsDNA titer from baseline to Day 56; a decrease in titer ≥ 35% was considered a positive response
Time Frame: baseline to Day 56
Population: The number of participants whose anti-dsDNA antibody titer decreased by ≥ 35% from baseline to Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Study With the Simon Two-Stage Trial Design
Number analyzed (Participants) | 10
Participants | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 84- 84 days
Description: Adverse events were assessed systematically by regular investigator assessments and regular laboratory testing.
Arm/Group | Open-label Study With the Simon Two-Stage Trial Design
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Study With the Simon Two-Stage Trial Design (N=15)
Abscess (Musculoskeletal and connective tissue disorders) | 1 (1) — right knee abscess culture + for proteus mirabilis.
Pyrexia (Immune system disorders) | 1 (1) — Admitted to the hospital with fever to 102, tachycardia and rash; all attributed to a lupus flare.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Study With the Simon Two-Stage Trial Design (N=15)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Abscess (Infections and infestations) | 2 (2)
Alopecia (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hepatic Enzyme increased (Hepatobiliary disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lupus Flare (Immune system disorders) | 1 (1)
Lymphadentiis (Infections and infestations) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Oropharyngeal pain (Infections and infestations) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (Immune system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper Respiratory tract infection (Infections and infestations) | 3 (3)
Viral Infection (Infections and infestations) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT02066311/Prot_SAP_000.pdf